CLINICAL TRIAL: NCT04168918
Title: Efficacy of a Group Psychological Intervention in Reducing Self-Stigma Among Outpatients at the Psychiatric Hospital: A Randomized Controlled Trial
Brief Title: Effectiveness of a Group Psychological Intervention in Reducing Self-stigma Among Patients With Mental Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Most participants did not complete the post-intervention questionnaire
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Shani Venner, Postgraduate student, The University of The West Indies
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 191002-A
Record Dates: First submitted 2019-11-14; First posted 2019-11-19 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Self-stigma; Self Efficacy; Quality of Life

STUDY DESIGN:
Intervention Model Description: Fifty per cent receive psychological intervention and fifty per cent receive treatment-as-usual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Psychological Intervention (Experimental): One topic will be discussed at each of the six sessions using some principles from cognitive behavioral therapy and psychoeducation.
  Interventions: Behavioral: Group psychological Intervention
- Treatment-as-usual (No Intervention): Participants will receive their usual care which involves being seen by a mental health professional (psychologist, psychiatrist/resident in psychiatry, or mental health nurse).

INTERVENTIONS:
Behavioral: Group psychological Intervention — There will be 6 sessions covering 6 topics (Understanding mental disorders, Self-stigma, Social support, Substance use and mental illness, Self-help strategies, Available mental health services). Each session will begin with welcoming, reviewing what was done in the last session and home assignments (where applicable), question-guided discussion, lecture, group sharing and home assignment
  Arms: Group Psychological Intervention

SUMMARY:
At the Psychiatric Hospital, there are limited mental health professionals to offer the standard of care that is expected at a psychiatric institution. Psychotherapy is most affected. However, there are mental health professionals in training and long waiting times before clients are seen, which provides an opportunity for an intervention to be carried out. The purpose of the study therefore, is to determine whether a group psychological intervention can primarily reduce self-stigma among outpatients at the Psychiatric Hospital. The intervention's effects on self-efficacy and quality of life will also be assessed.

DETAILED DESCRIPTION:
Study population: outpatients in the Outpatient Department at The Psychiatric Hospital

Target population: clients with two-weekly appointments

Procedures for recruitment and consent

Participants will be chosen using available lists of persons who come to clinic on a two-weekly basis on four(4) days of the week (every day except the day the Principal Investigator is responsible for conducting clinic), for two consecutive weeks. Twenty-six will be chosen each day (for eight (8) days) and randomized to intervention and treatment-as-usual (Thirteen (13) persons to each group). Participants will be selected based on the inclusion and exclusion criteria and consent will be obtained.

Randomization will be carried out by Stata 14

Sample size

Using the means and standard deviations for the Internalized Stigma of Mental Illness Inventory (ISMI) used in a randomized controlled trial and Stata 14 for sample size calculation, the sample size recommended is eighty-four (84) with forty-two (42) per group. This will give a power (for the study) of eighty per cent (80%).

However, the aim will be two-hundred and eight (208) clients based on the following:

* Target population: two-hundred and fifty (250). Approximately twenty-five (25) patients come to clinic daily, most of whom come on a two-weekly basis. Therefore, this will allow eighty-three per cent (83%) of the population to be part of the study.
* Maximum number of persons in a group- thirteen (13)
* Maximum number of groups that can be held before clinic begins- one (1)
* Time for thesis
* Taking into account that persons may not be willing to participate and so aiming to include as many persons as possible

Method

There will be six (6) sessions covering six (6) topics. One topic will be covered at each session. Sessions will last sixty (60) to ninety (90) minutes.

Data collection

- Administration of the ISMI, the General self-efficacy scale and World Health Organization (WHO)5 Well Being Index and a questionnaire to the intervention and control groups before the intervention and after the intervention. This will be done by a health professional not related to the study.

Permission was obtained from producer of ISMI. WHO5 Well-Being Index is free to use and General self-efficacy scale does not require permission, once referenced.

All three scales have been found to be valid and reliable.

* A pilot study on 26 persons will be conducted to test the questionnaire and scales.
* To ensure accurate completion of questionnaire and scales by each participant, each item will be read and explained before participants asked to select answer. Questions on clarification will be encouraged.Time will also be given after, for participants to read through answers if needed. Additionally, when collecting questionnaires and scales, the mental health professional will scan through to ensure all questions answered.

Questionnaires and scales will be identified using participants' record numbers to facilitate verification of information such as whether medications or health care provider changed during the course of the intervention.

Statistical analyses

* Summary statistics
* Regression analysis of endpoint score adjusting baseline score and looking at the difference between the intervention and treatment-as-usual groups.

Intention to treat analysis will be used.

- Software to be used: Stata 14 Missing entries will be included in the analysis Data handling and record keeping

Questionnaires kept in secure room for at least five (5) years

ELIGIBILITY:
Inclusion Criteria:

* Attend clinic every 2 weeks
* Willingness to attend all sessions

Exclusion Criteria:

* Cognitive impairment that limits the participant from understanding material and answering questions

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Change in self-stigma | From enrollment to the end of intervention at 12 weeks
  Mean Change from Baseline in scores on the Internalized Stigma of Mental Illness Inventory (ISMI) after 6 sessions Each item is scored 1-4 (1=strongly disagree;4=strongly agree), yielding a total between 29 and 116. Higher scores indicate greater self-stigma.

SECONDARY OUTCOMES:
Change in self-efficacy: General self-efficacy scale | From enrollment to the end of intervention at 12 weeks
  Mean Change from Baseline in scores on the General self-efficacy scale after 6 sessions Each item is scored 1-4 (1=not true at all; 4=exactly true) yielding a total between 10 and 40. Higher scores indicate more self-efficacy
Change in quality of life: WHO5 Well Being Index | From enrollment to the end of intervention at 12 weeks
  Mean Change from Baseline in scores on the WHO5 Well Being Index after 6 sessions Each item is scored 0-5 (0=at no time; 5=all of the time) yielding between 0 and 25. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Shani KM Venner, MBBS,MPH, Principal Investigator — University of the West Indies-Cave Hill Campus
Locations (1):
- The Psychiatric Hospital, Bridgetown, Barbados

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cuhadar D, Cam MO. Effectiveness of psychoeducation in reducing internalized stigmatization in patients with bipolar disorder. Arch Psychiatr Nurs. 2014 Feb;28(1):62-6. doi: 10.1016/j.apnu.2013.10.008. Epub 2013 Oct 28. PMID 24506989
- [Background] Schwarzer R, Jerusalem M. Generalized Self-Efficacy scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs (pp. 35-37). Windsor, UK: NFER-NELSON, 1995
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Chang CC, Wu TH, Chen CY, Wang JD, Lin CY. Psychometric evaluation of the internalized stigma of mental illness scale for patients with mental illnesses: measurement invariance across time. PLoS One. 2014 Jun 2;9(6):e98767. doi: 10.1371/journal.pone.0098767. eCollection 2014. PMID 24887440